CLINICAL TRIAL: NCT03719079
Title: The Nanowear Wearable Heart Failure Management System Multiple Sensor Algorithm Development and Validation Trial
Brief Title: Nanowear Heart Failure Management Multi-sensor Algorithm
Acronym: Nanosense
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanowear Inc. (Industry)
Collaborators: Milton S. Hershey Medical Center (Other); Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Other Study IDs: NWCT18-SS-001
Record Dates: First submitted 2018-10-23; First posted 2018-10-25 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Heart Failure
Keywords: Fluid decompensation; Non-invasive Multi-parameter monitoring; Multi-parameter algorithm; Heart Rate Variability; Thoracic impedance; Heart Sounds; Respiration; Posture; Activity; Tidal Volume; Stroke Volume
MeSH Terms: conditions — Heart Failure; Respiratory Aspiration; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Heart Failure Patients: Patients with primary diagnosis as heart failure
  Interventions: Device: SimpleSENSE

INTERVENTIONS:
Device: SimpleSENSE — The Nanosense study is observational only. No interventions will be triggered by the SimpleSense device

SUMMARY:
The NanoSense study is a multi-center, prospective, non-randomized, observational, feasibility, non-significant risk study. The NanoSense study will enroll up to 500 subjects in up to 10 centers in order to collect data which includes at least 150 heart failure hospitalizations in participating subjects.The duration of the NanoSense study is expected to be 2 years. The study device is the Wearable Congestive Heart Failure Management System (WCHFS, also known as SimpleSENSE)

DETAILED DESCRIPTION:
NanoSense is a data collection study to develop a multi-sensor algorithm to predict worsening Heart Failure (HF). Subjects who meet the eligibility criteria and agree to participate in the study will enter the informed consent process in which the subject will be informed about the research study, the voluntary nature of the research and all attendant risks and benefits. Once the subject has been informed and all question answered, the subject will be asked to sign an informed consent document (approved by the local Institutional Review Board). At enrollment, data about subject demographics, cardiac disease history, and comorbidities will be collected. The subject vital signs, blood labs (as available; if an N-terminal pro b-type natriuretic peptide (NT-proBNP) is not available, one will be ordered to coincide with the next lab samples), HF medications and HF assessment measurements will be made and recorded. Subjects will be given a diary to record daily weights, diuretics changes, and weekly HF status. The subject will be fitted with a Nanowear Wearable Congestive Heart Failure System (WCHFS) and educated on the use of the system with attention to proper fit and changing or charging the battery daily depending on the type of battery used. Subjects who have a pacemaker or Implantable Cardioverter Defibrillator (ICD) will undergo pacemaker/ICD interrogation while wearing the device to assure that there are no electrical signals detected that may interfere with pacemaker or ICD function.

The subjects will be asked to wear the device for approximately 12 hours daily including 2 hours prior to sleep and 2 hours after awakening. The follow-up period will be 90 days. At visit 2, the clinical assessment will be repeated and recorded. The device will be retrieved from the subject. In the event that a subject is unable to travel to the investigator's site, the subject will be asked to mail the device back to the sponsor with use of a prepaid mailing package that will be delivered to the subject. Data may be obtained by phone if the subject is unable or unwilling to return for visit 2.

A final contact will be made to the subject at 30 days following visit 2 to determine whether there were any adverse effects that were not previously recognized that may be related to their participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent
* Male or female over the age of 18 years
* The patient is either hospitalized with a primary diagnosis of acute or was discharged with a primary diagnosis of acute heart failure within 2 weeks prior to enrollment
* NYHA functional class II-IV at time of enrollment

Exclusion Criteria:

* Subject unwilling or unable to comply with wearing the Nanowear Congestive Heart Failure Management System 12 hours daily for up to 90 days.
* Subjects who are limited by angina.
* Severe aortic stenosis.
* Subjects who are hemodynamically unstable requiring support with intravenous vasoactive medications or mechanical circulatory support
* Symptomatic ventricular arrhythmias within the past 6 months.
* Subjects who are pregnant will be excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects of legal age to give informed consent who are currently or recently hospitalized with a primary diagnosis of heart failure
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-08-21 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Multi-parameter algorithm | 90 days per patient and till 100 Heart Failure events are observed overall.
  The primary objective of the study is to develop and validate a multi-parameter algorithm for the detection of heart failure prior to a HF event. For the purpose of this study, a heart failure event will be defined as a hospitalization with a primary diagnosis of heart failure.

SECONDARY OUTCOMES:
Exploratory comparison of signals from device to NT-proBNP | 90 days per patient and till 100 Heart Failure events are observed overall.
  Exploratory information will be used to compare the signals obtained from the device to the severity of heart failure as measured by clinical evaluation (NYHA functional class and physical examination) and NT-proBNP

CONTACTS AND LOCATIONS:
Overall Officials: John P Boehmer, M.D., Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States